CLINICAL TRIAL: NCT01960647
Title: Phase III FREERIDE STUDY Freeway Randomized Angioplasty Study
Brief Title: FREERIDE STUDY, Freeway Paclitaxel Coated Balloon Catheter to Treat Peripheral Artery Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eurocor GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eur-003
Record Dates: First submitted 2013-09-30; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uncoated PTA balloon catheter (Other): Dilatation with uncoated PTA balloon catheter
  Interventions: Device: Percutaneous transluminal angioplasty with uncoated balloon
- Freeway Paclitaxel balloon catheter (Active Comparator): Dilatation with Freeway Paclitaxel (3 µg/mm2) coated balloon catheter
  Interventions: Device: Percutaneous transluminal angioplasty with Paclitaxel balloon

INTERVENTIONS:
Device: Percutaneous transluminal angioplasty with uncoated balloon
  Arms: Uncoated PTA balloon catheter
Device: Percutaneous transluminal angioplasty with Paclitaxel balloon
  Arms: Freeway Paclitaxel balloon catheter

SUMMARY:
The primary objective of this prospective, Randomized, Controlled, Multicentre, Open Study is to investigate the inhibition of restenosis by the Paclitaxel-eluting Percutaneous transluminal angioplasty (PTA) balloon Freeway versus PTA alone in the treatment of de-novo occluded, stenotic or reoccluded, restenotic superficial femoral (SFA) or popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female (> 18 years of age) with symptomatic ischemia, requiring treatment of SFA or PI segment ( 2-5 of Rutherford classification)
* Single and/or multiple de novo occluded, stenotic or reoccluded, restenotic lesion(s) of > 70% , ≤ 15 cm in total length and vessel diameter ≥ 4mm and ≤ 7mm (by visual estimation).
* Patient provides a signed informed consent and complies with the follow up visits
* Successful wire crossing of lesion
* At least one patent (less than 50% stenosis) tibioperoneal run-off vessel

Exclusion Criteria:

* Gastrointestinal bleeding or coagulopathy contraindicating use of anti-platelet therapy
* Known intolerance contraindications to study medications and contrast agents, non-controllable with medication.
* Patient actively participating in another device or drug study
* History of hemorrhagic stroke within 3 months
* Previous or planned surgical or intervention procedure within 30 days of index procedure
* Significant untreated inflow disease or no normal arterial segment proximal of lesion in which duplex ultrasound velocity ratios can be measured
* Acute or sub-acute thrombus in target vessel
* Use of adjunctive therapies (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon)
* Patients with in-stent restenosis or prior surgery of the target lesion
* Patients with abdominal aortic, iliaca or popliteal aneurysm (AAA) with ≥ 4cm diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically driven target lesion revascularization | 6 months

SECONDARY OUTCOMES:
Technical success | Baseline
Clinical success | Baseline
Procedural success | Baseline
Ankle Brachial index improvement | 6, 12, 24 months
Change in Rutherford classification | 6, 12, 24 months
Walking improvement | 6, 12 ,24 months
Rate of minor and major complications | 6,12, 24 months
Rate of target lesion revascularization | 12, 24 months
Late lumen loss | 6 months
Patency rate | 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Ludwig Schulte, Prof. PhD, Principal Investigator — Ev. Krankenhaus Königin Elisabeth Herzberge. Berlin
Locations (17):
- Medical University, Graz, Austria
- Angiografia De Occidente, Cali, Colombia
- Germany (8):
  - Ev. Krankenhaus Königin Elisabeth Herzberge, Berlin, State of Berlin
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Berlin-Gefäßzentrum, Berlin
  - Klinikum Links der Weser, Bremen
  - Krankenhaus Dresden-Friedrichstadt, Dresden
  - Medical University, Leipzig
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tuebingen, Tübingen
- Semmelweis Universitíy, Budapest, Hungary
- Italy (5):
  - Policlinico Abano Terme, Abano Terme
  - Maria Cecilia Hospital, Cotignola
  - Casa di Cura Privata Montevergine S.p.a., Mercogliano
  - San Giovanni Battista "Molinette", Torino
  - San Giovanni Bosco Hospital, Torino
- Hospital Universitario de Donostia, Donostia / San Sebastian, Spain